CLINICAL TRIAL: NCT00429884
Title: Studies of Disorders and Mechanisms Related to Atrial Fibrillation Before and After DC-Conversion: Polysomnography, Heart Rate Variability and 24h Holter.
Brief Title: Studies of Disorders and Mechanisms Related to Atrial Fibrillation Before and After DC-Conversion.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Other Study IDs: 05-027M
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate if breathing disorders are related to atrial fibrillation and if it is possible to predict recurrence of atrial fibrillation after DC-conversion by changes in heart rate variability and 24 hour ECG.

ELIGIBILITY:
Inclusion Criteria:

* persistent atrial fibrillation
* scheduled for electrical cardioversion

Exclusion Criteria:

* known obstructive sleep apnea

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Steen M Jensen, MD, PhD, Principal Investigator — Heart Centre, Umeå University Hospital; Niklas G Höglund, MD, Principal Investigator — Heart Centre, Umeå University Hospital; Karl Franklin, MD, PhD, Principal Investigator — Umeå University Hospital
Locations (1):
- Heart Centre, Umeå University Hospital, Umeå, Sweden

REFERENCES:
- [Derived] Hoglund N, Sahlin C, Kesek M, Jensen SM, Franklin KA. Cardioversion of atrial fibrillation does not affect obstructive sleep apnea. Ups J Med Sci. 2017 Jun;122(2):114-118. doi: 10.1080/03009734.2017.1291545. Epub 2017 Mar 14. PMID 28291376